CLINICAL TRIAL: NCT03094013
Title: Psychosocial Factors of Burn Related Injuries and Perceived Gaps in Service Delivery During the Rehabilitation Period: A Mixed Methods Study
Brief Title: Psychosocial Factors of Burn Related Injuries and Perceived Gaps in Service Delivery
Status: Terminated | Type: Observational
Why Stopped: PI moved. Unable to recruit
Sponsor: St. Louis University (Other)
Collaborators: Mercy Research (Other)
Responsible Party: Sponsor
Other Study IDs: 944614; eRS 20227 (Other: St. Louis U)
Record Dates: First submitted 2017-02-02; First posted 2017-03-29 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Burns; Psychological
Keywords: psycho-social factors, psychological symptoms
MeSH Terms: conditions — Burns | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — Assessment

SUMMARY:
This study will utilize a mixed methods design featuring quantitative assessment of symptoms in conjunction with collecting in-depth qualitative data. In this study, perceived stress, mental health symptoms and behaviors and other variables will be used to test how they will influence the daily functioning and service utilization for adolescent and adult burn related injury patients at Mercy Hospital St. Louis Burn Center. The data gathered in the interviews will explore these constructs in-depth for the participants.

DETAILED DESCRIPTION:
Background:

Survivors of burn injury can experience a broad spectrum of physical and psychological outcomes depending on the burn severity (Esselman, 2007; Fauerbach et al., 2007). Strides in research have been made to further our understanding of burn related injuries, however, there are gaps in the literature concerning the areas of prevention, intervention, and improving outcomes for psychosocial adjustment post-burn, and a fractious and varied approach to the measurement of psychosocial adjustment (Attoe & Pounds-Cornish, 2015). Two major research areas have been identified as priority areas in burn research: further understanding psychosocial factors associated with burn related injuries and intervention related research (Fauerbach, Pruzindky, & Saxe, 2007; Attoe & Pounds-Cornish, 2015). Attoe & Pounds-Cornish (2015) identified the following constructs as warranting further study: depression anxiety disorders, phobias, substance abuse, sexuality, body image, peer support, post-traumatic growth, social support, active coping, sleep problems, bullying. Fauerbach, Pruzindky, & Saxe (2007) added that the role of length of hospital stay, personality, burn characteristics, and time since burn on return to work, work changes, and work satisfaction are also important factors to study.

There is, without question, an important bridge to be built between our emerging understanding of the psychosocial needs among burn survivors and the offering of hope through intervention (Fauerbach, Pruzindky, & Saxe, 2007). The first step to ensure that interventions are effective is to identify and assess which services and interventions are available, utilization of these services, patient satisfactions of services, measured outcomes, degree of compliance, facilitators and barriers to psychosocial interventions, impact of psychological and psychological stressors on outcomes, and gaps in services. Having a greater understanding of the psychosocial factors and needs among burn survivors has the potential to impact how services are developed, implemented, and utilized.

Research Objectives and Purpose:

The two research questions guiding this study are:

1. What are the psychological factors impacting burn related injury survivors?
2. What is the relationship between psychosocial factors for burn related injury survivors, discharge readiness, and service utilization?

This proposed study aims to:

1. Assess psychosocial symptoms, behaviors, and adjustment post-burn in adolescents, adults, and family members; and
2. Conduct a needs assessment related to post-burn services utilization, perception of service quality and service need, and facilitators and barriers to service delivery and utilization.

Research Methods:

Study design:

This study will utilize a mixed methods design featuring quantitative assessment of symptoms in conjunction with collection of in-depth qualitative data. A convergent parallel mixed methods design will be used, in which qualitative and quantitative data will be collected in parallel, analyzed separately, and then merged. In this study, perceived stress, mental health symptoms and behaviors and other variables will be used to test how they will influence the daily functioning and service utilization for adolescent an adult burn related injury patients. The data gathered in the interviews will explore these constructs in-depth for the participants.

Patients who are hospitalized due to a burn related injury who require skin grafts will be eligible to participate in this study. After it is determined by hospital staff that they are medically stabilized, hospital staff will give information to the patient about the study. This determination will be made with the clinical team (nurses, doctors, PAs, mental health professionals) and final determination will come from the clinical supervisor. If they agree to the initial pre-screening meeting, the PI will give detailed information about the study and will go through the consent procedure. Participation in this study is completely voluntary. Participation does not give patients any incentive related to care or services available.

Participation in the study will involve patients participating in comprehensive assessments during hospital stay, during discharge planning, and three times post-hospitalization. The goal is that 300 individuals participate in the comprehensive assessments over a two year period. Power analysis for cross-sectional data was conducted in Open Source Epidemiologic Statistics for Public Health to determine a sufficient sample size using an alpha of 0.05, a power of 0.80, a medium effect size (ρ = 0.30), and one tail (Faul et al., 2008). Based on the aforementioned assumptions, the desired sample size is 95 (utilizing data related to PTSD with a conservative 22% rate with outcome). A sample size of 300 will give sufficient power for analysis of factors that may have lower prevalence.

Data Collection for quantitative data:

1. Once enrolled in the study, the PI will collect the initial baseline assessment data from study participants during meetings. Sociodemographic data will include items such as age (at time of first assessment, while participant is still in the hospital), race and ethnicity, household income, perceived financial stability, marital status, and work and school related information. The baseline assessment includes discharge questions asked during the discharge process. The assessment instrument includes the following measures/assessment questions. The surveys will be completed interview style, with the PI marking answers to the questions. Data will be entered into Qualtrics, a secure online survey program.

   1. Relevant demographic information
   2. CFPB Financial Well-Being Scale Questionnaire
   3. Psychosocial Assessment
   4. Sleep - Wake Questionnaire (University of South Carolina)
   5. Perceived Stress Scale: This 10-item scale measures the perception of stress (Cohen, Kamarck, & Mermelstein, 1983).
   6. Burn's Depression Checklist
   7. Burn's Anxiety Inventory
   8. Rosenberg Self-Esteem Scale: A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self (Rosenberg, 1965).
   9. WHO Disability Assessment Schedule 2.0
   10. Satisfaction with Appearance Scale
   11. Sexual Distress Scale
   12. Adverse Childhood Experience Questionnaire
   13. PTSD Checklist for DSM-5 with Life Events Checklist: This 20-item self-report measure assesses the twenty DSM-5 symptoms of Post Traumatic Stress Disorder (Weathers, Litz, Keane, Palmieri, Marx, & Schnurr, 2013).
   14. Dissociative Subtype of PTSD Scale (DSPS): The DSPS is a 15-item measure that assesses lifetime and past-month (current) dissociative symptoms, including symptoms that define the DSM-5 definition of the dissociative subtype of PTSD (Wolf, Mitchell, Sadeh, Hein, Fuhrman, Pietrzak, & Miller, in press).
   15. Center for Epidemiological Studies Depression Scale for Children (CES-DC) (Faulstich, Carey, Ruggiero et al., 1986)
   16. Screen for Child Anxiety Related Disorders (SCARED) (Birmaher, Brent, Chiappetta, Bridge, Monga, & Baugher, 1999)
   17. UCLA PTSD Index for DSM (Adolescent version)
   18. Adolescent Dissociative Experiences Scale-II (A-DES) (Armstrong, Putnam, Carlson, Libero, & Smith, 1997)
   19. Discharge questions

       First meeting: during hospitalization and during discharge planning Demographic information (Adults, Adolescents, Parents) CFPB Financial Well-Being Scale Questionnaire (Adults, Parents) Psychosocial assessment (Adults, Adolescents, Parents) Sleep - Wake Questionnaire (Adults, Adolescents) Perceived Stress Scale (Adults, Adolescents) Burn's Depression Checklist (Adults) Burn's Anxiety Inventory (Adults) Rosenberg Self-Esteem Scale (Adults, Adolescents) WHO Disability Assessment Schedule 2.0 (Adults, Adolescents) Satisfaction with Appearance Scale (Adults, Adolescents) Sexual Distress Scale (Adults) Adverse Childhood Experience Questionnaire (Adults) PTSD Checklist for DSM-5 with Life Events Checklist (Adults) Dissociative Subtype of PTSD Scale (Adults) Center for Epidemiological Studies Depression Scale for Children (Adolescents) Screen for Child Anxiety Related Disorders (Adolescents) UCLA PTSD Index for DSM (Adolescent version) (Adolescents) Adolescent Dissociative Experiences Scale-II (Adolescents) Discharge questions (Adults, Adolescents, Parents) Second meeting: approximately 1 month post-discharge CFPB Financial Well-Being Scale Questionnaire (Adults, Parents) Psychosocial assessment (Adults, Adolescents, Parents) Sleep - Wake Questionnaire (Adults, Adolescents) Perceived Stress Scale (Adults, Adolescents) Burn's Depression Checklist (Adults) Burn's Anxiety Inventory (Adults) Rosenberg Self-Esteem Scale (Adults, Adolescents) WHO Disability Assessment Schedule 2.0 (Adults, Adolescents) Satisfaction with Appearance Scale (Adults, Adolescents) Sexual Distress Scale (Adults) PTSD Checklist for DSM-5 with Life Events Checklist (Adults) Dissociative Subtype of PTSD Scale (Adults) Center for Epidemiological Studies Depression Scale for Children (Adolescents) Screen for Child Anxiety Related Disorders (Adolescents) UCLA PTSD Index for DSM (Adolescent version) (Adolescents) Adolescent Dissociative Experiences Scale-II (Adolescents) Third meeting: approximately 6 months post-discharge CFPB Financial Well-Being Scale Questionnaire (Adults, Parents) Psychosocial assessment (Adults, Adolescents, Parents) Sleep - Wake Questionnaire (Adults, Adolescents) Perceived Stress Scale (Adults, Adolescents) Burn's Depression Checklist (Adults) Burn's Anxiety Inventory (Adults) Rosenberg Self-Esteem Scale (Adults, Adolescents) WHO Disability Assessment Schedule 2.0 (Adults, Adolescents) Satisfaction with Appearance Scale (Adults, Adolescents) Sexual Distress Scale (Adults) PTSD Checklist for DSM-5 with Life Events Checklist (Adults) Dissociative Subtype of PTSD Scale (Adults) Center for Epidemiological Studies Depression Scale for Children (Adolescents) Screen for Child Anxiety Related Disorders (Adolescents) UCLA PTSD Index for DSM (Adolescent version) (Adolescents) Adolescent Dissociative Experiences Scale-II (Adolescents) Fourth meeting: approximately 1 year post-discharge CFPB Financial Well-Being Scale Questionnaire (Adults, Parents) Psychosocial assessment (Adults, Adolescents, Parents) Sleep - Wake Questionnaire (Adults, Adolescents) Perceived Stress Scale (Adults, Adolescents) Burn's Depression Checklist (Adults) Burn's Anxiety Inventory (Adults) Rosenberg Self-Esteem Scale (Adults, Adolescents) WHO Disability Assessment Schedule 2.0 (Adults, Adolescents) Satisfaction with Appearance Scale (Adults, Adolescents) Sexual Distress Scale (Adults) PTSD Checklist for DSM-5 with Life Events Checklist (Adults) Dissociative Subtype of PTSD Scale (Adults) Center for Epidemiological Studies Depression Scale for Children (Adolescents) Screen for Child Anxiety Related Disorders (Adolescents) UCLA PTSD Index for DSM (Adolescent version) (Adolescents) Adolescent Dissociative Experiences Scale-II (Adolescents)
2. One month post-discharge, the PI will again collect the assessment data.
3. Six months post-discharge, the PI will again collect the assessment data.
4. One year post-discharge, the PI will collect that last assessment data.

Data Collection for qualitative data:

The investigators will utilize a sample of participants (both adults and adolescents) for the in-depth interviews. The investigators will randomly select a subset of participants from the larger sample, who may be stratified by age, gender, work-related vs. non work-related injuries, or other injury characteristics. This depends on the participant data available. The investigators plan to include approximately 50 participants for the qualitative in-depth interviews at approximately 6 months from discharge from the hospital. Once data is stratified, individuals who have consented to participate in the qualitative portion will be randomized and asked to participate in the full interview.

In depth interviews will be conducted with 25 participants each grant year (total of 50 participants). The interviews will consist of more in depth questions related to functioning, symptoms, stressors, services available, services utilized, financial and community resources, gaps in service delivery, perceptions of discharge preparation, satisfaction with services received, emotional and physical preparedness during recovery stages, and short and long term worries and goals.

Interviews will be recorded and transcribed by a professional transcription service (no identifiable data will be included in recordings).

Data Collection from hospital staff:

The investigators will use a survey to ask hospital staff about their perceptions of hospital-based service utilization. The goal is for 15 staff members to complete either the on-line or in person survey. Data collected from hospital staff will be entered into Qualtrics (for in person interviews) and directly entered into Qualtrics online.

Study Participants:

The investigators anticipate that 300 participants will be enrolled in the study over a two year period.

Inclusion Criteria for Adults and Adolescents:

* Ages: 16 years and older
* Males and females
* Individuals with burn related injuries requiring a skin graft and in the hospital long enough to complete the first assessment.

Exclusion Criteria

• Individuals with burn related injuries, but who do not receive skin grafts. Individuals who are physically or mentally unable to give consent for participation.

Inclusion Criteria for Mercy Hospital Staff:

* Currently working in the St. Louis Burn Center in Mercy Hospital
* Males and females

Recruitment, Informed Consent, and Financial Information:

When patients in the Burn Center are physically stabilized, the hospital staff will inform patients of the study. They will have the option to participate in a pre-screening meeting where the PI goes through the study and consent information.

Consent will take place once hospital staff determine that the patient is physically, medically stabilized, before discharge. With input from other hospital staff, the Physician Assistant will make the final determination if the patient is ready to be asked about their participation in this study. The PA will use both written materials and the script to give information to potential participants. Potential participants will be given time to consider their participation while in the hospital, with understanding that participation would start before discharge.

Both consent from parents and assent from individuals will be required for any adolescents in the study. They will have full access to mental health services during their hospital stay. They will also be given information about community mental health services available. If any current abuse or neglect is reported, the study PI will follow reporting guidelines to ensure the safety of the child.

The youngest children will be 16 and 17 years old and will be asked for the assent for participation. Participants can stop their participation at any time and can skip any questions. Questions do not go beyond typical psychological examinations. Participants will have access to mental health services.

Hospital staff will be notified about the study during weekly staff meetings and via email. They will directly contact the PI if they would like to participate in the study. After signing consent forms, they will decide if they would like to participate in the online survey or in the in person interview meeting.

Risk Assessment:

Participants may feel discomfort while answering questions related to personal information and symptoms, especially if they have negative memories associated with the topics or experiences.

Participants will have access to in-hospital psychological and counseling services. After discharge, they will have access to community resources that provide mental health services. In addition, participants will be informed that they can stop their participation at any time and they can skip any questions that make them uncomfortable.

Due to the nature of some of the questions in the questionnaires, the PI collecting data will continually check-in with study participants and monitor any symptoms, feelings, and thoughts that come up during the meetings or interviews. Because of the sensitive nature, the meetings will take place in person, so the PI collecting the data can visibly monitor participant responses. In addition, between instruments, the PI will ask the participant if she/he is able to continue and if she/he is experiencing any distress. If a participant discloses intention to harm self or others, the PI will follow Missouri state reporting laws. If a participant reports distress and/or strong emotions that they feel that they cannot self-regulate or regulate through grounding and relaxation techniques utilized by the PI, the PI and participant will decide the best course of action. If the meeting is held outside of Mercy Hospital, this may include calling 911 or accompanying to the nearest hospital. The PI will also have a list of community mental health resources that she will give to study participants and assist participants to make appointments, when appropriate. While in the hospital, the participant can be referred to psychological and counseling services, if she/he is not already actively receiving services. The PI will ensure that the hospital clinical staff members are aware of any reported distress (with participant permission).

Potential Benefits

There is no known direct benefit to individual participants.

This research study is significant in multiple ways. This study involves two major research areas that have been identified as priority areas: further understanding of psychosocial factors associated with burn related injuries and intervention related research. The proposal includes an in depth analysis of multiple psychosocial factors that have been identified as needing further study. The study also involves a needs assessment related to intervention strategies currently utilized at Mercy Hospital St. Louis Burn Center and has the potential to impact service delivery and utilization by identifying factors related to successes, facilitators and barriers, perceived gaps in service, and perceptions in discharge preparation. The results of this study can guide policy, practice, and future research both at a local and national level.

Understanding the psychosocial factors related to burn related injury survivors is important to improve current services for individuals and their families and develop needed services. Identifying facilitators and barriers also aids in ensuring that individuals and their families have access to these services. Ultimately, participation in the study adds to the small knowledge base that seeks to alleviate psychological and emotional distress that individuals and their families experience.

Data Confidentiality and Participant Privacy:

Participants will be assigned an ID number that will be utilized on all documents. The ID number and name key will be held on the PI's computer, which will be password protected. Any health information utilized for the study will be entered using only the ID number. Only the PIs will have access to the data obtained in this study. Electronic data will be password protected. Paper data (only containing ID numbers) will be stored in a locked file cabinet in a locked office. Data collected from hospital staff will be entered into Qualtrics (for in person interviews) and directly entered into Qualtrics online. Therefore no information from the hospital staff will be kept at Mercy Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with burn related injuries requiring a skin graft and in the hospital long enough to complete the first assessment.

Exclusion Criteria:

* Individuals with burn related injuries, but who do not receive skin grafts.
* Individuals who are physically or mentally unable to give consent for participation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 300 individuals with burn related injuries requiring a skin graft and in the hospital long enough to complete the first assessment, receiving in-patient care at Mercy Hospital Burn Center.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | baseline (during hospitalization)
  stress levels (adults, adolescents)
Burn's Depression Checklist | baseline (during hospitalization)
  depressive symptoms (adults)
Burn's Anxiety Inventory | baseline (during hospitalization)
  anxiety symptoms (adults)
PTSD Checklist for DSM-5 with Life Events Checklist, Adverse Childhood Experiences Questionnaire, Dissociative Subtype of PTSD Scale | baseline (during hospitalization)
  trauma symptoms (adults)
Center for Epidemiological Studies Depression Scale for Children | baseline (during hospitalization)
  depressive symptoms (adolescents)
Screen for Child Anxiety Related Disorders | baseline (during hospitalization)
  anxiety symptoms (adolescents)
UCLA PTSD Index for DSM (Adolescent version), Adolescent Dissociative Experiences Scale-II | baseline (during hospitalization)
  trauma symptoms (adolescents)
Discharge readiness questions | discharge (approx 2-6 weeks after initial hospitalization)
  adults and adolescents
Perceived Stress Scale | approximately 1 month post-hospitalization (after discharge)
  stress levels (adults, adolescents)
Burn's Depression Checklist | approximately 1 month post-hospitalization
  depressive symptoms (adults)
Burn's Anxiety Inventory | approximately 1 month post-hospitalization
  anxiety symptoms (adults)
PTSD Checklist for DSM-5 with Life Events Checklist, Adverse Childhood Experiences Questionnaire, Dissociative Subtype of PTSD Scale | approximately 1 month post-hospitalization
  trauma symptoms (adults)
Center for Epidemiological Studies Depression Scale for Children | approximately 1 month post-hospitalization
  depressive symptoms (adolescents)
Screen for Child Anxiety Related Disorders | approximately 1 month post-hospitalization
  anxiety symptoms (adolescents)
UCLA PTSD Index for DSM (Adolescent version), Adolescent Dissociative Experiences Scale-II | approximately 1 month post-hospitalization
  trauma symptoms (adolescents)
Perceived Stress Scale | approximately 6 months post-hospitalization
  stress levels (adults, adolescents)
Burn's Depression Checklist | approximately 6 months post-hospitalization
  depressive symptoms (adults)
Burn's Anxiety Inventory | approximately 6 months post-hospitalization
  anxiety symptoms (adults)
PTSD Checklist for DSM-5 with Life Events Checklist, Adverse Childhood Experiences Questionnaire, Dissociative Subtype of PTSD Scale | approximately 6 months post-hospitalization
  trauma symptoms (adults)
Center for Epidemiological Studies Depression Scale for Children | approximately 6 months post-hospitalization
  depressive symptoms (adolescents)
Screen for Child Anxiety Related Disorders | approximately 6 months post-hospitalization
  anxiety symptoms (adolescents)
UCLA PTSD Index for DSM (Adolescent version), Adolescent Dissociative Experiences Scale-II | approximately 6 months post-hospitalization
  trauma symptoms (adolescents)
Perceived Stress Scale | approximately 1 year post- hospitalization
  stress levels (adults, adolescents)
Burn's Depression Checklist | approximately 1 year post- hospitalization
  depressive symptoms (adults)
Burn's Anxiety Inventory | approximately 1 year post- hospitalization
  anxiety symptoms (adults)
PTSD Checklist for DSM-5 with Life Events Checklist, Adverse Childhood Experiences Questionnaire, Dissociative Subtype of PTSD Scale | approximately 1 year post- hospitalization
  trauma symptoms (adults)
Center for Epidemiological Studies Depression Scale for Children | approximately 1 year post- hospitalization
  depressive symptoms (adolescents)
Screen for Child Anxiety Related Disorders | approximately 1 year post- hospitalization
  anxiety symptoms (adolescents)
UCLA PTSD Index for DSM (Adolescent version), Adolescent Dissociative Experiences Scale-II | approximately 1 year post- hospitalization
  trauma symptoms (adolescents)

SECONDARY OUTCOMES:
CFPB Financial Well-Being Scale Questionnaire | baseline (during hospitalization)
  financial well-being (adults and parents)
CFPB Financial Well-Being Scale Questionnaire | approximately 1 month post-hospitalization (after discharge)
  financial well-being (adults and parents)
CFPB Financial Well-Being Scale Questionnaire | approximately 6 months post-hospitalization
  financial well-being (adults and parents)
CFPB Financial Well-Being Scale Questionnaire | approximately 1 year post-hospitalization
  financial well-being (adults and parents)
Sleep - Wake Questionnaire | baseline (during hospitalization)
  sleep (adults and adolescents)
Sleep - Wake Questionnaire | approximately 1 month post-hospitalization
  sleep (adults and adolescents)
Sleep - Wake Questionnaire | approximately 6 months post-hospitalization
  sleep (adults and adolescents)
Sleep - Wake Questionnaire | approximately 1 year post-hospitalization
  sleep (adults and adolescents)
Rosenberg Self-Esteem Scale | baseline (during hospitalization)
  self-esteem (adults and adolescents
Rosenberg Self-Esteem Scale | approximately 1 month post-hospitalization
  self-esteem (adults and adolescents
Rosenberg Self-Esteem Scale | approximately 6 months post-hospitalization
  self-esteem (adults and adolescents
Rosenberg Self-Esteem Scale | approximately 1 year post-hospitalization
  self-esteem (adults and adolescents
WHO Disability Assessment Schedule 2.0 | during hospitalization
  physical functioning (adults and adolescents)
WHO Disability Assessment Schedule 2.0 | approximately 1 month post-hospitalization
  physical functioning (adults and adolescents)
WHO Disability Assessment Schedule 2.0 | approximately 6 months post-hospitalization
  physical functioning (adults and adolescents)
WHO Disability Assessment Schedule 2.0 | approximately 1 year post-hospitalization
  physical functioning (adults and adolescents)
Satisfaction with Appearance Scale | during hospitalization
  physical appearance satisfaction (adults and adolescents)
Satisfaction with Appearance Scale | approximately 1 month post-hospitalization
  physical appearance satisfaction (adults and adolescents)
Satisfaction with Appearance Scale | approximately 6 months post-hospitalization
  physical appearance satisfaction (adults and adolescents)
Satisfaction with Appearance Scale | approximately 1 year post-hospitalization
  physical appearance satisfaction (adults and adolescents)
Sexual Distress Scale | during hospitalization
  (adults)
Sexual Distress Scale | approximately 1 month post-hospitalization
  (adults)
Sexual Distress Scale | approximately 6 months post-hospitalization
  (adults)
Sexual Distress Scale | approximately 1 year post-hospitalization
  (adults)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Fearn, PhD, Study Director — Director-School of Social Work
Locations (1):
- Mercy Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attoe C, Pounds-Cornish E. Psychosocial adjustment following burns: An integrative literature review. Burns. 2015 Nov;41(7):1375-84. doi: 10.1016/j.burns.2015.02.020. Epub 2015 Sep 8. PMID 26359733
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Beck, A. T., Steer, R.A., & Garbin, M.G. (1988) Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clinical Psychology Review, 8(1), 77-100.
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Esselman PC. Burn rehabilitation: an overview. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S3-6. doi: 10.1016/j.apmr.2007.09.020. PMID 18036978
- [Background] Fauerbach JA, Pruzinsky T, Saxe GN. Psychological health and function after burn injury: setting research priorities. J Burn Care Res. 2007 Jul-Aug;28(4):587-92. doi: 10.1097/BCR.0B013E318093E470. No abstract available. PMID 17514031
- [Background] Wolf EJ, Mitchell KS, Sadeh N, Hein C, Fuhrman I, Pietrzak RH, Miller MW. The Dissociative Subtype of PTSD Scale: Initial Evaluation in a National Sample of Trauma-Exposed Veterans. Assessment. 2017 Jun;24(4):503-516. doi: 10.1177/1073191115615212. Epub 2015 Nov 23. PMID 26603115
- [Background] Wortmann JH, Jordan AH, Weathers FW, Resick PA, Dondanville KA, Hall-Clark B, Foa EB, Young-McCaughan S, Yarvis JS, Hembree EA, Mintz J, Peterson AL, Litz BT. Psychometric analysis of the PTSD Checklist-5 (PCL-5) among treatment-seeking military service members. Psychol Assess. 2016 Nov;28(11):1392-1403. doi: 10.1037/pas0000260. Epub 2016 Jan 11. PMID 26751087